CLINICAL TRIAL: NCT00856167
Title: TCM for TMD: A Multi-Site Whole Systems Trial
Brief Title: Traditional Chinese Medicine (TCM) for Temporomandibular Dysfunction (TMD): A Whole Systems Multi-site Trial
Acronym: TCM-TMD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-0289-01; U01AT002570 (NIH)
Record Dates: First submitted 2009-03-03; First posted 2009-03-05 (Estimated); Results first posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2022-06

CONDITIONS: Temporomandibular Dysfunction
Keywords: temporomandibular dysfunction; TMD; TMJ; Traditional Chinese Medicine; TCM
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Medicine, Chinese Traditional; Self Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional Chinese Medicine (Active Comparator): Whole systems traditional Chinese medicine, including herbal formulas, acupuncture, tuna (Chinese massage), lifestyle recommendations
  Interventions: Combination Product: Traditional Chinese Medicine
- Self-care (Active Comparator): Self-care for TMD developed by Dworkin, LeResche et al.
  Interventions: Behavioral: Self-care for TMD

INTERVENTIONS:
Combination Product: Traditional Chinese Medicine — Whole systems traditional Chinese medicine, including individually tailored herbal formulas based on a formulary, acupuncture (based on individual TCM diagnoses), tuna (Chinese massage), lifestyle recommendations
  Arms: Traditional Chinese Medicine
Behavioral: Self-care for TMD — a 5-session 8 hour intervention targeting TMD knowledge, stretching and exercises, stress reduction, lifestyle modification
  Arms: Self-care

SUMMARY:
This study sought to evaluate the benefits of different combinations of a Self Care program, involving individually targeted education and support, plus Traditional Chinese Medicine, in terms of patients' experience and outcomes in short-term follow-up (8 weeks, reported here) and long-term follow-up (18-months). The study seeks to evaluate the benefits and drawbacks of different patterns of stepped care, which means different levels of care depending on patients' responses at various time-points in the study, which might be used by clinicians treating in the future.

DETAILED DESCRIPTION:
Studies of temporomandibular disorders (TMD) have shown that chronic pain in the temporomandibular joint (TMJ) and/or masticatory muscles affects more than 10% of adults at any one time and that one-third of adults will experience TMD over their lifespan (Von Korff et al. 1988). TMD includes a wide range of symptoms: facial pain, jaw-joint pain, headaches, earaches, dizziness, masticatory musculature hypertrophy, limited mouth opening, closed or open lock on the TMJ, abnormal occlusal wear, clicking or popping sounds in the jaw joint, and other complaints (NIH 1996). Although the etiology is poorly understood, longitudinal data suggest that TMD is an enduring, recurrent condition and a resistant problem for many (Dworkin et al. 1992a; Dworkin et al. 1989; Moss 1982; Gale 1978), and it affects individuals in all socioeconomic and ethnic groups (Smith & Syrop 1994). In a study of TMD patients in Kaiser Permanente Northwest (KPNW) in 1990-1995, the mean age was 40.5 years, and 80% of the patients were female. TMD subjects used 1.6 times the services of other health plan members (White 2001).

The Research Diagnostic Criteria for TMD (RDC/TMD) proposed by Dworkin et al. (Dworkin & LeResche 1992b) uses a dual axis system for diagnosing and classifying TMD patients. Axis I assigns physical diagnoses of the most commonly occurring masticatory muscle and/or TMJ disorders (arthralgia, arthritis, and arthroses of the TMJ). Axis II assesses behavioral, psychological and psychosocial factors; functional mandibular limitations; psychological distress, including depression; and Graded Scale of Chronic Pain (GCP) (Von Korff et al. 1992). The RDC/TMD criteria for Axes I and II have been used in numerous clinical research studies around the world (Ohrbach & Dworkin 1998; List et al. 1996; Rudy et al. 1995; Garofalo & Wesley 1998; Yap et al. 2002). An NIH-supported international consortium of RDC/TMD clinical researchers has been established to foster multinational studies of TMD using as their core the RDC/TMD standardized methods and criteria (http://www.rdc-tmdinternational.org/). The RDC/TMD has been suggested as a model system for the diagnosis and assessment of all chronic pain conditions (Garofolo & Wesley 1997; Dworkin, Sherman et al. 2002). The RDC/TMD is being used in this study for the primary endpoint.

Epidemiological studies of TMD have focused on estimating prevalence and describing characteristics of persons with and without the condition (Carlsson & LeResche 1995). In more than 75% of the studies reviewed, TMD was not adequately defined. Epidemiologic and clinical studies of TMD confirm its fundamental status as a chronic pain problem (Bell 1986; Fricton et al. 1987; Dworkin et al. 1992a). Yap et al. (2003) found that about 39% of TMD patients also are depressed, and 55% exhibit elevated levels of somatization. Similarly, Lee et al. (1995) found that TMD patients frequently present ear pain, neck pain, shoulder pain, headaches, and previous head or neck trauma.

Despite a number of temporomandibular joint pain clinical trials, no approach has been found to persistently and significantly reduce the severity and disability of this condition. The investigators' recent phase II RCT (n=110 women) showed that Traditional Chinese Medicine (TCM), including acupuncture and herbs, was comparable to or better than comprehensive specialty usual care in reducing pain, and better in improving disability. The improvements did not persist, however, once TCM treatment ended. The investigators hypothesize that this may have been due in part to their lack of education in self-care management. Thus, when their pain returned, they knew of no other option than returning to their TCM practitioner which was not permitted under the protocol. This suggests that the appropriate way to incorporate TCM into TMD care should include a self-care component for all participants. This proposal tests TCM versus self- care management (SC) in a realistic manner that is consistent with an integrative, stepped care strategy, one that begins with a minimal self-care intervention (one session) and increases the intensity in relation to patient needs. After period 1 allocation to TCM or self-care, participants not already on TCM will be allocated to self-care or TCM if period 2 if continued treatment is warranted. This study design is more clinically meaningful than a customary two-group randomization, which does not consider patient outcomes (see study Schema below).

The investigators propose a two-site (Tucson and Portland) phase II trial (n=150) that will evaluate the potential short-term pain benefits of TCM. The study hypothesis is that in the two-step clinical allocation model, TCM participants will experience more characteristic facial pain reduction than those who receive only self-care. The investigators will expand the patient population beyond their previous study to include both men and women, as well as individuals who have received previous TMD care (not TCM) and continue to experience TMD pain.

ELIGIBILITY:
Inclusion Criteria:

* TMD as diagnosed according to the Research Diagnostic Criteria-TMD by a trained dentist;
* worst facial pain greater than 5 out of 10.

Exclusion Criteria:

* prior surgery for TMD;
* life-threatening illnesses;
* conditions that would prevent participation in trial including consumption of Chinese herbs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2006-10 (Actual); Primary Completion 2010-01 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Ritenbaugh, PhD, MPH, Principal Investigator — U of Arizona

REFERENCES:
- [Result] Ritenbaugh C, Hammerschlag R, Dworkin SF, Aickin MG, Mist SD, Elder CR, Harris RE. Comparative effectiveness of traditional Chinese medicine and psychosocial care in the treatment of temporomandibular disorders-associated chronic facial pain. J Pain. 2012 Nov;13(11):1075-89. doi: 10.1016/j.jpain.2012.08.002. Epub 2012 Oct 9. PMID 23059454
- [Result] Elder C, Ritenbaugh C, Aickin M, Hammerschlag R, Dworkin S, Mist S, Harris RE. Reductions in pain medication use associated with traditional Chinese medicine for chronic pain. Perm J. 2012 Summer;16(3):18-23. doi: 10.7812/TPP/12.967. PMID 23012594

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study took place in Tucson, Arizona, and Portland, Oregon, recruited through newspaper advertisements, and various email list-serves. In Tucson, there was also an active community outreach component to enhance the recruitment of minorities. All individuals responded to our call center in Tucson using a toll-free number. Recruitment began October 1, 2006 and ended September 1, 2007.
Pre-assignment Details: In the 1st period, 79 subjects were allocated to TCM (39) or SC (40). 36 TCM subjects completed the 1st period; all were removed from the allocation group for the 2nd period per study plan. 35 SC subjects completed the 1st period. 29 were allocated to TCM (15) or SC (14) for the 2nd period; 6 were removed from the allocation group due to subject choice or insufficient pain. 56 additional subjects were allocated to TCM (27) or SC (29) for the 2nd period. 135 subjects total were allocated.
Groups:
- Traditional Chinese Medicine - Period 1; Traditional Chinese Medicine - Period 2: Whole systems traditional Chinese medicine, including individually tailored herbal formulas, acupuncture, tuna (Chinese massage), lifestyle recommendations
  TCM: whole system Traditional Chinese Medicine, including acupuncture, herbs, tuina, lifestyle counseling
- Self-care - Period 1; Self Care - Period 2: Self-care for TMD developed by Dworkin, LeResche et al.
  Self-care for TMD: a 5-session 8 hour intervention targeting TMD knowledge, stretching and exercises, stress reduction, lifestyle modification
Period: Period 1
Arm/Group | Traditional Chinese Medicine - Period 1 | Self-care - Period 1 | Traditional Chinese Medicine - Period 2 | Self Care - Period 2
Started | 39 | 40 | 0 | 0
Completed | 36 | 35 | 0 | 0
Not Completed | 3 | 5 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0
Period: Period 2
Arm/Group | Traditional Chinese Medicine - Period 1 | Self-care - Period 1 | Traditional Chinese Medicine - Period 2 | Self Care - Period 2
Started | 0 | 0 | 42 | 43
Completed | 0 | 0 | 37 | 38
Not Completed | 0 | 0 | 5 | 5
Not completed — Lost to Follow-up | 0 | 0 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Self Care - Period 1; Self Care - Period 2: Self-care for TMD developed by Dworkin, LeResche et al. Self-care for TMD: a 5-session 8 hour intervention targeting TMD knowledge, stretching and exercises, stress reduction, lifestyle modification
- Total: Total of all reporting groups
Arm/Group | Traditional Chinese Medicine - Period 1 | Self Care - Period 1 | Traditional Chinese Medicine - Period 2 | Self Care - Period 2 | Total
Number analyzed (Participants) | 39 | 40 | 42 | 43 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: In the 1st period, 79 subjects were allocated to TCM (39) or SC (40). 36 TCM subjects completed the 1st period; all were removed from the allocation group for the 2nd period per study plan. 35 SC subjects completed the 1st period. 29 were allocated to TCM (15) or SC (14) for the 2nd period; 6 were removed from the allocation group due to subject choice or insufficient pain. 56 additional subjects were allocated to TCM (27) or SC (29) for the 2nd period. 135 subjects total were allocated.
  years
    Period 1: number analyzed (Participants) | 39 | 40 | 0 | 0 | 79
    Period 1 | 42.9 (13.0) | 42.3 (13.5) |  |  | 42.6 (13.3)
    Period 2: number analyzed (Participants) | 0 | 0 | 42 | 43 | 85
    Period 2 |  |  | 43.6 (12.0) | 43.7 (12.4) | 43.65 (12.20)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: In the 1st period, 79 subjects were allocated to TCM (39) or SC (40). 36 TCM subjects completed the 1st period; all were removed from the allocation group for the 2nd period per study plan. 35 SC subjects completed the 1st period. 29 were allocated to TCM (15) or SC (14) for the 2nd period; 6 were removed from the allocation group due to subject choice or insufficient pain. 56 additional subjects were allocated to TCM (27) or SC (29) for the 2nd period. 135 subjects total were allocated.
  Participants
    Period 1: number analyzed (Participants) | 39 | 40 | 0 | 0 | 79
    Period 1: Female | 34 | 34 |  |  | 68
    Period 1: Male | 5 | 6 |  |  | 11
    Period 2: number analyzed (Participants) | 0 | 0 | 42 | 43 | 85
    Period 2: Female |  |  | 37 | 37 | 74
    Period 2: Male |  |  | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: In the 1st period, 79 subjects were allocated to TCM (39) or SC (40). 36 TCM subjects completed the 1st period; all were removed from the allocation group for the 2nd period per study plan. 35 SC subjects completed the 1st period. 29 were allocated to TCM (15) or SC (14) for the 2nd period; 6 were removed from the allocation group due to subject choice or insufficient pain. 56 additional subjects were allocated to TCM (27) or SC (29) for the 2nd period. 135 subjects total were allocated.
  Participants
    Period 1: number analyzed (Participants) | 39 | 40 | 0 | 0 | 79
    Period 1: Hispanic or Latino | 4 | 4 |  |  | 8
    Period 1: Not Hispanic or Latino | 33 | 34 |  |  | 67
    Period 1: Unknown or Not Reported | 2 | 2 |  |  | 4
    Period 2: number analyzed (Participants) | 0 | 0 | 42 | 43 | 85
    Period 2: Hispanic or Latino |  |  | 5 | 5 | 10
    Period 2: Not Hispanic or Latino |  |  | 35 | 38 | 73
    Period 2: Unknown or Not Reported |  |  | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: In the 1st period, 79 subjects were allocated to TCM (39) or SC (40). 36 TCM subjects completed the 1st period; all were removed from the allocation group for the 2nd period per study plan. 35 SC subjects completed the 1st period. 29 were allocated to TCM (15) or SC (14) for the 2nd period; 6 were removed from the allocation group due to subject choice or insufficient pain. 56 additional subjects were allocated to TCM (27) or SC (29) for the 2nd period. 135 subjects total were allocated.
  Participants
    Period 1: number analyzed (Participants) | 39 | 40 | 0 | 0 | 79
    Period 1: American Indian or Alaska Native | 0 | 0 |  |  | 0
    Period 1: Asian | 1 | 0 |  |  | 1
    Period 1: Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
    Period 1: Black or African American | 1 | 1 |  |  | 2
    Period 1: White | 33 | 33 |  |  | 66
    Period 1: More than one race | 1 | 1 |  |  | 2
    Period 1: Unknown or Not Reported | 3 | 5 |  |  | 8
    Period 2: number analyzed (Participants) | 0 | 0 | 42 | 43 | 85
    Period 2: American Indian or Alaska Native |  |  | 0 | 0 | 0
    Period 2: Asian |  |  | 0 | 0 | 0
    Period 2: Native Hawaiian or Other Pacific Islander |  |  | 0 | 0 | 0
    Period 2: Black or African American |  |  | 0 | 0 | 0
    Period 2: White |  |  | 35 | 37 | 72
    Period 2: More than one race |  |  | 0 | 0 | 0
    Period 2: Unknown or Not Reported |  |  | 7 | 6 | 13
Region of Enrollment [Number; unit: participants] — Period 1 participants living in United States Population: In the 1st period, 79 subjects were allocated to TCM (39) or SC (40). 36 TCM subjects completed the 1st period; all were removed from the allocation group for the 2nd period per study plan. 35 SC subjects completed the 1st period. 29 were allocated to TCM (15) or SC (14) for the 2nd period; 6 were removed from the allocation group due to subject choice or insufficient pain. 56 additional subjects were allocated to TCM (27) or SC (29) for the 2nd period. 135 subjects total were allocated.
  participants
    United States: number analyzed (Participants) | 39 | 40 | 0 | 0 | 79
    United States | 39 | 40 |  |  | 79
Region of Enrollment [Number; unit: participants] — Period 2 participants living in the United States Population: In the 1st period, 79 subjects were allocated to TCM (39) or SC (40). 36 TCM subjects completed the 1st period; all were removed from the allocation group for the 2nd period per study plan. 35 SC subjects completed the 1st period. 29 were allocated to TCM (15) or SC (14) for the 2nd period; 6 were removed from the allocation group due to subject choice or insufficient pain. 56 additional subjects were allocated to TCM (27) or SC (29) for the 2nd period. 135 subjects total were allocated.
  participants
    United States: number analyzed (Participants) | 0 | 0 | 42 | 43 | 85
    United States |  |  | 42 | 43 | 85

OUTCOME MEASURES:

1. Primary Outcome: Characteristic Facial Pain Score
Description: The Characteristic Facial Pain (CFP) score is a mean of participant-reported worst pain over the previous two weeks, average pain when having pain over the previous two weeks, and current pain, reported on a 0-10 VAS scale where 0 means no pain and 10 means worst possible pain.
Time Frame: Beginning of each treatment period, end of each treatment period (8 weeks later)
Population: In the 1st period, 79 subjects were allocated to TCM (39) or SC (40). 36 TCM subjects completed the 1st period; all were removed from the allocation group for the 2nd period per study plan. 35 SC subjects completed the 1st period. 29 were allocated to TCM (15) or SC (14) for the 2nd period; 6 were removed from the allocation group due to subject choice or insufficient pain. 56 additional subjects were allocated to TCM (27) or SC (29) for the 2nd period. 135 subjects total were allocated.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Traditional Chinese Medicine - Period 1 | Self-care - Period 1 | Traditional Chinese Medicine - Period 2 | Self Care - Period 2
Number analyzed (Participants) | 36 | 35 | 37 | 38
units on a scale
  Period 1 - Pre-treatment: number analyzed (Participants) | 36 | 35 | 0 | 0
  Period 1 - Pre-treatment | 6.52 (1.24) | 6.55 (1.40) |  |
  Period 1 - Post-treatment: number analyzed (Participants) | 36 | 35 | 0 | 0
  Period 1 - Post-treatment | 5.11 (1.70) | 5.47 (2.09) |  |
  Period 2 - Pre-treatment: number analyzed (Participants) | 0 | 0 | 37 | 38
  Period 2 - Pre-treatment |  |  | 5.34 (1.54) | 5.22 (1.43)
  Period 2 - Post-treatment: number analyzed (Participants) | 0 | 0 | 37 | 38
  Period 2 - Post-treatment |  |  | 4.44 (1.70) | 4.93 (1.54)
Statistical Analysis 1: Comparison: Traditional Chinese Medicine - Period 1 vs Self-care - Period 1 vs Traditional Chinese Medicine - Period 2 vs Self Care - Period 2; Participants were allocated to one of the two treatments in order to balance baseline CFP, a depression score, age, gender, and site (Tucson or Portland); Test type: Superiority; p = 0.020, Regression, Linear — Regression coefficient of TCM indicator variable, with change in CFP as the outcome, and controlling for start of treatment values: CFP, depression, gender, age, site; Regression coefficient = -0.60; Since some participants could appear in both the 1st and 2nd period, the regression included random effects to account for correlation between measures on the same person. In the 1st period, participants could either be allocated to TCM or SC, or if their pain scores were below 5, simply assigned to continuing self-care. Comparisons from this period were only between the allocated TCM and SC groups. In the 2nd period, those allocated or assigned to SC in the 1st period could be allocated to TCM or SC, or again assigned to continuing SC if their pain scores were too low. Comparisons from this period were only between the allocated TCM and SC groups

ADVERSE EVENTS:
Time Frame: Adverse events were solicited at every regular data collection to six months beyond completion of any treatment; all practitioners had forms to use for any adverse event at a treatment session.
Description: Symptoms were monitored per DSMB to locate possible harms, using a checklist of 24 that might be from herbs, acupuncture, lifestyle changes, recommended self-care, and as new; severity; treatment-related; change since previous. Response protocols were in place. Each DSMB reviewed patterns x intervention. Ppts reported use of emergency rooms or hospital admissions since prior query. Every "yes" required follow-up. All final decisions were by medical directors consensus with PI /DSMB concurrence.
Groups:
- Traditional Chinese Medicine - Period 1; Traditional Chinese Medicine - Period 2: Whole systems traditional Chinese medicine, including herbal formulas, acupuncture, tuna (Chinese massage), lifestyle recommendations
  Traditional Chinese Medicine: Whole systems traditional Chinese medicine, including individually tailored herbal formulas based on a formulary, acupuncture (based on individual TCM diagnoses), tuna (Chinese massage), lifestyle recommendations
Arm/Group | Traditional Chinese Medicine - Period 1 | Self-care | Traditional Chinese Medicine - Period 2 | Self Care - Period 2
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/40 | 0/43 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/40 | 0/43 | 0/42
Other Adverse Events (participants affected / at risk) | 1/39 | 0/40 | 0/43 | 0/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Traditional Chinese Medicine - Period 1 (N=39) | Self-care (N=40) | Traditional Chinese Medicine - Period 2 (N=43) | Self Care - Period 2 (N=42)
Ear cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | NA | NA — Ear cellulitis due to acupuncture needles in a woman who had intermittent ear cellulitis prior to the acupuncture. In response to this, practitioners queried participants about cellulitis history before administering acupuncture.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No